CLINICAL TRIAL: NCT02881463
Title: Prehabilitation Physical Activity: Relationship With Muscle Function, Postural Stability and Postoperative Recovery in Persons With Osteoarthritis
Brief Title: Prehabilitation Physical Activity in Persons With Osteoarthritis
Acronym: PrehabOA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Helena Gapeyeva, Research Fellow, Md, PhD, University of Tartu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 218/T-16
Record Dates: First submitted 2016-06-16; First posted 2016-08-29 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Home Exercise Program (Experimental): 8- week therapeutical exercise program performing at home for women with knee joint osteoarthritis
  Interventions: Other: therapeutical exercises

INTERVENTIONS:
Other: therapeutical exercises — Participants of experimental group performs daily an 8-week home therapeutical exercise program. Exercises are periodized by weeks (1-8 weeks). The aim of program is the leg muscle strengthening using an elastic band (Thera-Band, System of Progressive Exercise, USA), body balance training, and leg muscle stretching.

SUMMARY:
Knee joint osteoarthritis (OA) reduces functional mobility and performance of daily tasks such as rising from a chair. Therefore interventions aimed at improving muscle strength and sit-to-stand task performance are very important for these patients. The effect of exercise programs, including home exercise programs (HEP), on muscle strength, joint pain and function is well known and widely researched, yet not many studies have investigated the effect of an HEP on electromyographic activity (EMG) of muscles when performing everyday tasks, such as rising from and sitting on a chair. The aim of this study was to investigate effect of prehabilitation in women with severe knee joint OA scheduled for knee joint arthroplasty (TKA).

ELIGIBILITY:
Inclusion Criteria:

* For OA patients: patients with severe knee joint OA undergoing unilateral total knee arthroplasty (TKA)
* for controls: pain of joints more than 20/100 mm by VAS

Exclusion Criteria:

For both groups:

* previous total joint arthroplasty of lower limbs
* other musculoskeletal, neurological and cardiovascular diseases
* any diseases affecting balance and coordination.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Muscle electromyographic (EMG) activity | up to 12 months
  Electromyographic (EMG) activity of thigh muscles during gait and sit to stand task (amplitude, mV)

SECONDARY OUTCOMES:
Knee joint pain intensity | up to 12 months
  Self-reported knee joint pain intensity measured by visual-analogue scale (VAS) (in mm: "0 mm" - no pain and "100 mm" - extreme pain)
Knee joint function | up to 12 months
  Self-reported functional status measured by Knee Injury and Osteoarthritis Outcome Score (KOOS) - Symptoms, Pain, Daily Living Activity, Sport and Recreational Activity. Quality of Life. Maximum is 100 points (complains are absent) and minimum is 0 points (extreme complains)
Sit to Stand test | up to 12 months
  five time Sit to Stand test from standard chair (s)
Mobility test | up to 12 months
  Timed Up and Go test, 3-m plus return 3-m walking test (s)
Leg muscles strength | up to 12 months
  strength of leg extensor muscles (N)
Body balance | up to 12 months
  Body postural sway measuring during standing using Kistler force plate (Switzerland) (mm), eyes open and eyes closed
Gait pattern | up to 12 months
  Gait kinematic characteristics measurement using three-dimensional movement analysis system and six optoelectronic cameras (BTS S.p.A. Italy) - joint angles (degrees)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Gapeyeva, MD, PhD, Principal Investigator — University of Tartu, Faculty of Medicine, Estonia

IPD SHARING:
Plan to Share IPD: Undecided